CLINICAL TRIAL: NCT00542542
Title: Prospective Randomized Clinical Trial to Evaluate the Use of Paravertebral Blocks in Reconstructive Breast Surgery
Brief Title: Evaluate the Use of Paravertebral Block in Reconstructive Breast Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2006-0961; NCI-2012-01557 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2007-10-10; First posted 2007-10-11 (Estimated); Results first posted 2015-04-13 (Estimated); Last update posted 2015-04-13 (Estimated); Status verified 2015-03

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Reconstructive Surgery; Paravertebral Block; Anesthesia; Propofol; Fentanyl; Ropivacaine; Midazolam
MeSH Terms: conditions — Breast Neoplasms | interventions — Propofol; Fentanyl; Ropivacaine; Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Paravertebral Block + General Anesthesia (Active Comparator): Group 1: Paravertebral Block + General Anesthesia (Ropivacaine)
  Interventions: Procedure: Paravertebral Block; Drug: Ropivacaine
- General Anesthesia Alone (Active Comparator): Group 2: General Anesthesia Alone (Propofol, Midazolam, Fentanyl)
  Interventions: Drug: Propofol; Drug: Fentanyl; Drug: Midazolam

INTERVENTIONS:
Procedure: Paravertebral Block — Paravertebral block given as a bolus injection into the paravertebral space.
  Arms: Paravertebral Block + General Anesthesia
Drug: Propofol — 2-2.5 mg/kg IV over 1-4 hours during surgery.
  Arms: General Anesthesia Alone
Drug: Fentanyl — 50-250 mcg IV over 1-4 hours during surgery.
  Arms: General Anesthesia Alone
Drug: Ropivacaine — Ropivacaine given by injection into the paravertebral space along the spinal canal.
  Arms: Paravertebral Block + General Anesthesia
Drug: Midazolam — 0.08 mg/kg IV over 1-4 hours during the surgery.
  Arms: General Anesthesia Alone

SUMMARY:
Primary Objective:

To determine whether the use of a paravertebral block in patients undergoing reconstructive surgery for breast cancer results in decreased immediate post-operative pain compared with patients having only general anesthesia.

Secondary Objectives:

1. To determine whether the use of a paravertebral block in patients undergoing reconstructive surgery for breast cancer results in decreased post-operative pain in the first 24 hours after surgery compared with patients having only general anesthesia.
2. To determine whether the use of a paravertebral block in patients undergoing reconstructive surgery for breast cancer results in decreased post-operative nausea and vomiting in the first 24 hours as compared with patients having only general anesthesia.
3. To determine whether the use of a paravertebral block in patients undergoing reconstructive surgery for breast cancer results in a decreased length of hospital stay compared with patients having only general anesthesia.

DETAILED DESCRIPTION:
Paravertebral Blocks and General Anesthesia The use of a paravertebral block involves injecting local anesthesia (a numbing medicine) into the patient's back to numb specific areas (the breast[s] for this study) for surgery.

General anesthesia is medicine that is used to put patients to sleep so that there is no feeling of pain.

Study Groups:

If you are found to be eligible to take part in this study, you will be randomly assigned (as in the toss of a coin) to 1 of 2 groups. You will have an equal (50/50) chance of being assigned to either group.

Participants in one group will receive a paravertebral block (the local anesthetic ropivacaine) plus general anesthesia.

Participants in the other group will receive general anesthesia (propofol, desflurane, and fentanyl) without a paravertebral block.

Drug Administration:

If you are assigned to receive the paravertebral block plus general anesthesia, you will have a paravertebral block placed just before surgery begins. Ropivacaine will be given by injection into the paravertebral space along the spinal canal.

If you are assigned to receive general anesthesia without a paravertebral block, you will be given propofol, desflurane, and fentanyl by vein over 1-4 hours during surgery.

Participants in both groups will receive promethazine, famotidine, and dexamethasone at the start of surgery to help decrease or eliminate nausea and vomiting that may occur after surgery.

Follow-up:

After your surgery is complete, before you leave the hospital, you will have the following evaluations:

* You will be asked how you are feeling so that the study doctor can determine how much medication you may need for pain and nausea as well as how long your hospital stay may need to be. You may be given fentanyl and dilaudid for pain and ondansetron and promethazine for nausea.
* You will also be asked about your satisfaction with the anesthesia. You will be asked these questions within the first hour, between 1 and 3 hours, and between 3 and 6 hours after surgery. Once you are discharged from the hospital, study staff will contact you by phone or talk with you when you return for a visit (at 18 -22 hours and 1 week after surgery) to ask these questions. It will take about 3-5 minutes to ask these questions each time.

Length of Study:

Your participation in this study will be over after the 1 week follow-up telephone call.

This is an investigational study. Paravertebral blocks and general anesthesia are FDA approved and commercially available. Up to 89 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients that consent to participate
2. Patients undergoing reconstructive breast surgery either in combination with oncologic surgery or alone
3. Patients that are female
4. Patients that are over the age of 18
5. Patients on anti-coagulants or other blood thinning medications will be eligible for inclusion if they stop taking these medications for at least the time specified below prior to date of surgery: Low molecular weight heparin must stop at least 36 hours prior to surgery. Coumadin must stop at least 5 days prior to surgery. Aspirin, Plavix and NSAIDs must stop at least 7 days prior to surgery.

Exclusion Criteria:

1. Patients on chronic anti-emetics (ie. chronic= more than once every two days for greater than 2 weeks)
2. Patients on chronic pain medication (ie. chronic= more than once every two days for greater than 2 weeks) excluding Aspirin, acetaminophen and NSAID's
3. Patients with BMI<20 or >40
4. Patients that are pregnant
5. Patients with chronic pain syndromes.
6. Patients with hypersensitivity to ropivacaine/amide-type anesthetics should be excluded from this trial as this would be a contraindication

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2007-09; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Farzin Goravanchi, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: September 10, 2007 to February 28, 2011. All recruitment done at The University of Texas (UT) MD Anderson Cancer Center.
Pre-assignment Details: Of the 89 participants enrolled, one participant was excluded prior to group assignment.
Groups:
- Group 1: Paravertebral Block + General Anesthesia: Paravertebral Block + General Anesthesia (Ropivacaine)
  Paravertebral Block: Paravertebral block given as a bolus injection into the paravertebral space.
  Ropivacaine: Ropivacaine given by injection into the paravertebral space along the spinal canal.
- Group 2: General Anesthesia Alone: General Anesthesia Alone (Propofol, Midazolam, Fentanyl)
  Propofol: 2-2.5 mg/kg IV over 1-4 hours during surgery.
  Fentanyl: 50-250 mcg IV over 1-4 hours during surgery.
  Midazolam: 0.08 mg/kg IV over 1-4 hours during the surgery.
Period: Overall Study
Arm/Group | Group 1: Paravertebral Block + General Anesthesia | Group 2: General Anesthesia Alone
Started | 44 | 44
Completed | 44 | 44
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: One participant was removed prior to study randomization.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: Paravertebral Block + General Anesthesia | Group 2: General Anesthesia Alone | Total
Number analyzed (Participants) | 44 | 44 | 88
Age, Continuous [Median (Full Range); unit: years] | 49 [27 to 75] | 51 [27 to 81] | 51 [27 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 44 | 88
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 44 | 44 | 88

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With No Pain Immediately After Surgery
Description: Pain assessed using a verbal numeric rating scale (NRS) scored by numeric integers, with scores of 0-10 where 0 is no pain and 10 is the worst pain. Pain evaluated within the first hour, between 1 - 3 hours, between 3 - 6 hours post-operatively. Additional reporting planned for following morning (18 - 24 hours post-operatively).
Time Frame: Starting immediately after surgery, every 2 hours till the 6th hour following surgery
Population: Analysis was not possible from data collected due to reporting inconsistencies.
Arm/Group | Group 1: Paravertebral Block + General Anesthesia | Group 2: General Anesthesia Alone
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse Event Reporting was from baseline to end of study involvement, approximately 21 days. Overall active study period from December 03, 2007 to March 05 2011.
Arm/Group | Group 1: Paravertebral Block + General Anesthesia | Group 2: General Anesthesia Alone
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/44
Other Adverse Events (participants affected / at risk) | 0/44 | 0/44

LIMITATIONS AND CAVEATS:
The study completed with measurement reporting issues (inconsistencies) leading to uninterpretable data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No